CLINICAL TRIAL: NCT02623855
Title: Stay Healthy In Nature Everyday: a Randomized Controlled Trial of the Effect of Family Nature Outings on Stress and Physical Inactivity in a Low Income Population
Brief Title: Stay Healthy In Nature Everyday: Family Nature Outings in a Low Income Population
Acronym: SHINE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UCSF Benioff Children's Hospital Oakland (Other)
Collaborators: East Bay Regional Park District (Other); National Recreation and Park Association (Other); University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2015-042
Record Dates: First submitted 2015-11-24; First posted 2015-12-08 (Estimated); Results first posted 2019-02-18 (Actual); Last update posted 2020-11-30 (Actual); Status verified 2020-11

CONDITIONS: Stress, Psychological; Social Isolation; Physical Activity
Keywords: Parks; Well-being; Stress; Physical Activity; Nature; Greenspace
MeSH Terms: conditions — Stress, Psychological; Social Isolation; Motor Activity | interventions — Case Management

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Park prescription (Active Comparator): Park prescription, pedometry.
  Interventions: Behavioral: Park prescription; Device: Pedometry
- Park prescription and family outings (Experimental): Park prescription, pedometry, case management and 3 weekly family outings.
  Interventions: Behavioral: Family outings; Behavioral: Park prescription; Device: Pedometry; Behavioral: Case Management

INTERVENTIONS:
Behavioral: Family outings — Participants will be invited to three weekly outings to local parks, case management and support in getting to nature. Participants will be offered transportation to the outings and s meal at local nature destinations. Programming at the park will include a picnic and walk with nature exploration, and will be facilitated by park and clinic staff.
  Arms: Park prescription and family outings
Behavioral: Park prescription — Participants will receive a map of local parks, and the recommendation to be physically active outdoors three days a week in nature.
Device: Pedometry — Participants will record their daily pedometry.
Behavioral: Case Management — Participants will receive a phone call to list potential barriers to participating in nature outings, and will talk through solutions with an investigator. Participants will be offered assistance with transportation if necessary.
  Arms: Park prescription and family outings

SUMMARY:
The SHINE study is a randomized controlled study of the effect of a park-based family support group on multiple outcomes (including stress and physical activity) in a low income population.

DETAILED DESCRIPTION:
Despite mounting evidence that nature matters for human health, we are not aware of any prospective intervention trials looking at the use of nature as a health intervention. Like other protective factors, such as the presence of a caring adult, safe play places, greater stimulation, the presence of green-space in a child's life has been empirically linked to greater resilience. Nature has been proposed as a buffer to stress through several pathways: by providing a space for friends and families to gather (thereby increasing social support and improving family relationships), by increasing opportunities for physical activity, and by improving cognition. Research to date suggests that participation in outdoor activities facilitates a sense of connectedness to place. This sense of attachment may also provide a form of social support. Families served by Children's Hospital Oakland Primary Care Clinic experience high levels of stress. As a safety-net clinic, the primary care clinic serves a diverse set of patients, with a common thread of poverty. The Stay Healthy In Nature program was developed to encourage stress management skills through play and physical activity in parks. The program uses a combination of facilitated and independent outings into local parks to encourage sustained behavior change and measurable health benefits.

ELIGIBILITY:
Inclusion Criteria:

* Child must be 4 years and older, a patient in our clinic, physically able, available for follow up, able to answer questionnaire
* Caregiver must be 18 or older, legal guardian, physically able, able for follow up, able to answer questionnaire

Exclusion Criteria:

* Enrolled in a weight loss program, unable to be physically active, unable to give informed consent, unable to follow up for study duration.

Min Age: 4 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2015-07; Primary Completion 2016-09 (Actual); Study Completion 2017-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nooshin Razani, MD, MPH, Principal Investigator — UCSF Benioff Children's Hospital Oakland
Locations (1):
- UCSF Benioff Children's Hospital Oakland Primary Care Clinic, Oakland, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Razani N, Morshed S, Kohn MA, Wells NM, Thompson D, Alqassari M, Agodi A, Rutherford GW. Effect of park prescriptions with and without group visits to parks on stress reduction in low-income parents: SHINE randomized trial. PLoS One. 2018 Feb 15;13(2):e0192921. doi: 10.1371/journal.pone.0192921. eCollection 2018. PMID 29447248

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Park Prescription | Park Prescription and Family Outings
Started | 56 | 100
Completed | 46 | 84
Not Completed | 10 | 16

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Park Prescription | Park Prescription and Family Outings | Total
Number analyzed (Participants) | 56 | 100 | 156
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 28 | 50 | 78
  Between 18 and 65 years | 28 | 50 | 78
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 72 | 106
  Male | 22 | 28 | 50
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African-American | 39 | 59 | 98
  Non-Latino White | 1 | 5 | 6
  Latino | 4 | 21 | 25
  Other (Native American, Middle Eastern, API) | 12 | 17 | 29
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 56 | 100 | 156

OUTCOME MEASURES:

1. Primary Outcome: Change in Stress
Description: measured through the Perceived Stress Score10 (PSS10) over 0, 1 and 3 months. The PSS10 is a ten item, validated instrument which ranges from 0-40. Each item on the instrument is summed to create a total score. Higher values correspond with higher stress.
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Park Prescription | Park Prescription and Family Outings
Number analyzed (Participants) | 23 | 42
units on a scale | -1.48 [-4.55 to 1.60] | -1.83 [-3.42 to -0.25]
Statistical Analysis 1: Comparison: Park Prescription vs Park Prescription and Family Outings; The study is powered for our primary outcome, caregiver stress as measured by the 10-item perceived stress s score (PSS10). Normative data from population samples show a mean PSS10 score of 13.2 points with a standard deviation of 6.35 points and a within-subject correlation coefficient of 0.77 over 2 weeks.We powered the study to detect a three point difference in the change of the PSS10. This effect size is consistent with other estimates of a clinically significant change; Test type: Superiority — Our hypothesis was that park prescriptions with group visits would have a superior result than park prescriptions alone; p = 0.6099, t-test, 2 sided

2. Primary Outcome: Change in Stress
Description: measured through the Perceived Stress Score10 (PSS10), a ten item, validated instrument which ranges from 0-40.
Time Frame: 1 month
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Park Prescription | Park Prescription and Family Outings
Number analyzed (Participants) | 21 | 39
units on a scale | -2.81 [-6.51 to 0.89] | -1.90 [-3.70 to -0.89]

3. Secondary Outcome: Change in Park Visits Per Week
Description: Self-reported number of park visits in the last week, measured at 0, 1, and 3 months.
Time Frame: 1 month
Measure: Mean (95% Confidence Interval); unit: park visits/week
Arm/Group | Park Prescription | Park Prescription and Family Outings
Number analyzed (Participants) | 23 | 42
park visits/week | 1.81 [0.82 to 2.80] | 1.08 [0.24 to 1.92]
Statistical Analysis 1: Comparison: Park Prescription vs Park Prescription and Family Outings; Test type: Superiority; p = 0.0085, t-test, 2 sided

4. Secondary Outcome: Change in Minutes of Moderate Physical Activity Per Day
Description: Parents will report their physical activity in terms of minutes of moderate physical activity in the week before follow up at 0, 1, and 3 months out.
  Pedometers were also given to participants. Of note, because of poor follow through with returning pedometer data, this variable was not analyzed in the study results.
Time Frame: 3 months
Population: Minutes of moderate physical activity per average day in the week prior to follow up at 0, 1 and 3 months was measured. Below we list the mean within group change of minutes of moderate physical activity per day.
Measure: Mean (95% Confidence Interval); unit: minutes/day
Arm/Group | Park Prescription | Park Prescription and Family Outings
Number analyzed (Participants) | 78 | 78
minutes/day | 33.91 [8.20 to 59.62] | 18.58 [3.75 to 33.42]

5. Secondary Outcome: Change in Cortisol Level in Parents
Description: Salivary cortisol from parents
Time Frame: 3 months
Measure: Mean (95% Confidence Interval); unit: ug/dL
Arm/Group | Park Prescription | Park Prescription and Family Outings
Number analyzed (Participants) | 17 | 35
ug/dL | -0.01 [-0.04 to 0.03] | 0.01 [-0.07 to 0.09]
Statistical Analysis 1: Comparison: Park Prescription vs Park Prescription and Family Outings; Test type: Superiority; p = 0.1749, t-test, 2 sided

6. Secondary Outcome: Change in Minutes of Moderate Physical Activity Per Day
Description: Parents will report their physical activity in terms of minutes of moderate physical activity in the week before follow up at 0, 1months follow up.
  Pedometers were also given to participants. Of note, because of poor follow through with returning pedometer data, this variable was not analyzed in the study results.
Time Frame: 1 month
Population: as for outcome 4
Measure: Mean (95% Confidence Interval); unit: minutes/day
Arm/Group | Park Prescription | Park Prescription and Family Outings
Number analyzed (Participants) | 18 | 38
minutes/day | 20.72 [-4.96 to 46.41] | 30.76 [8.28 to 53.25]

7. Secondary Outcome: Change in Cortisol Level in Parents
Description: Salivary cortisol from parents
Time Frame: 1 month
Measure: Mean (95% Confidence Interval); unit: ug/dL
Arm/Group | Park Prescription | Park Prescription and Family Outings
Number analyzed (Participants) | 17 | 35
ug/dL | -0.01 [-0.04 to 0.03] | 0.01 [-0.07 to 0.09]

8. Secondary Outcome: Change in Park Visits Per Week
Description: Self-reported number of park visits in the last week, measured at 0, 1, and 3 months.
Time Frame: 3 month
Measure: Mean (95% Confidence Interval); unit: park visits/week
Arm/Group | Park Prescription | Park Prescription and Family Outings
Number analyzed (Participants) | 23 | 42
park visits/week | -1.48 [-4.55 to 1.60] | -1.83 [-3.42 to -0.25]

ADVERSE EVENTS:
Arm/Group | Park Prescription | Park Prescription and Family Outings
All-Cause Mortality (participants affected / at risk) | 0/28 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/28 | 0/50
Other Adverse Events (participants affected / at risk) | 0/28 | 0/50

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No